CLINICAL TRIAL: NCT06196593
Title: Visual Outcomes Following Bilateral Implantation of a Non-diffractive Wavefront-shaping Extended Depth of Focus Toric Intraocular Lens
Brief Title: Visual Outcomes Following Bilateral Implantation of the Vivity Toric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LEC Eye Centre (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Mun Wai Lee, Medical Director, LEC Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTLEC
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Cataract Senile; Intraocular Lens Complication
Keywords: cataract surgery; intraocular lens; non-diffractive extended depth of focus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All eyes (Experimental): All eyes implanted with AcrySof™ IQ Vivity™ Toric intraocular lens
  Interventions: Device: AcrySof™ IQ Vivity™ Toric intraocular lens

INTERVENTIONS:
Device: AcrySof™ IQ Vivity™ Toric intraocular lens — Uneventful phacoemulsification and implantation of IOL

SUMMARY:
The objective of this study was to evaluate the clinical and patient reported outcomes after bilateral implantation of the AcrySof™ IQ Vivity™ Toric intraocular lens.

DETAILED DESCRIPTION:
This is a prospective interventional case series of 30 patients who underwent cataract surgery and bilateral implantation of the AcrySof™ IQ Vivity™ Toric intraocular lens. This study is represented by an Asian cohort of patients and the study evaluations were focused not only on clinical visual outcomes but also on "real-life" patient reported outcomes such as dysphotopsias, spectacle independence and daily visual tasks all of which were measured at 1 month and up to 3 months postoperatively. The objective would be to provide insight into the performance of this intraocular lens in Asian patients.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* bilateral significant cataracts
* bilateral significant corneal astigmatism

Exclusion Criteria:

* previous refractive surgery
* amblyopia
* strabismus
* any ocular co-morbidity which could impact on final visual acuity
* pre-existing zonular weakness
* capsular instability or compromise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Binocular UDVA | 3 months
  Binocular Uncorrected Distance Visual Acuity
Binocular UIVA | 3 months
  Binocular Uncorrected Intermediate Visual Acuity
Binocular UNVA | 3 months
  Binocular Uncorrected Near Visual Acuity

SECONDARY OUTCOMES:
CDVA | 3 months
  Corrected Distance Visual Acuity
DCIVA | 3 months
  Distance Corrected Intermediate Visual Acuity
DCNVA | 3 months
  Distance Corrected Near Visual Acuity
MRSE | 3 months
  Mean Refractive Spherical Equivalent
Rotational Stability | 1 month
  Degree of rotation of intraocular lens
Binocular Defocus Curve | 3 months
  Measurement of the performance of the Intraocular lens at different distances
Contrast Sensitivity | 3 months
  Measurement of the contrast sensitivity after implantation with this intraocular lens
QUVID | 3 months
  Questionnaire on Visual Disturbances
VF-14 | 3 months
  Visual function 14 index of questions designed to assess difficulty performing daily visual tasks

CONTACTS AND LOCATIONS:
Locations (1):
- LEC Eye Centre, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-12-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT06196593/Prot_000.pdf